CLINICAL TRIAL: NCT07119463
Title: The Application and Effect of Goal-oriented Albumin Infusion in the Control of Postoperative Complications in Patients With Gastric Cancer - a Single-center Prospective Non- Randomized Controlled Study
Brief Title: Effect of Goal-Oriented Albumin Infusion on Postoperative Complication Management in Gastric Cancer Surgery
Acronym: GOAI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Yuchen Guo, Ph.D., Prof., The First Hospital of Jilin University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOAI
Record Dates: First submitted 2025-06-19; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Hypoalbuminemia; Postoperative Complications; Gastric Cancer
Keywords: Gastric Cancer; Postoperative Hypoalbuminemia; Albumin Infusion; Goal-Oriented Therapy; Postoperative Complications; Clavien-Dindo Classification; Nutritional Support
MeSH Terms: conditions — Postoperative Complications; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Albumin Threshold Group（25g/L）（LAT Group） (Experimental): Participants in this group will receive albumin infusion when serum albumin levels fall below 25 g/L during the postoperative period. The intervention aims to maintain serum albumin levels above this threshold to evaluate its impact on complications and recovery.
  Interventions: Drug: Human Serum Albumin Infusion for LAT Group
- High Albumin Threshold Group (30 g/L)(HAT Group) (Active Comparator): Participants in this group will receive albumin infusion when serum albumin levels fall below 30 g/L during the postoperative period. This group serves as the control to compare the effects of a higher albumin threshold on complications and recovery.
  Interventions: Drug: Human Serum Albumin Infusion for HAT Group

INTERVENTIONS:
Drug: Human Serum Albumin Infusion for LAT Group — Participants in this group will receive human serum albumin infusion when their serum albumin level falls below 25 g/L. The infusion is goal-oriented, with the aim of maintaining albumin levels above 25 g/L during the postoperative period. The dose is calculated based on the albumin deficit and patient weight to ensure optimal therapeutic effect.
  Arms: Low Albumin Threshold Group（25g/L）（LAT Group）
Drug: Human Serum Albumin Infusion for HAT Group — Participants in this group will receive human serum albumin infusion when their serum albumin level falls below 30 g/L. The intervention aims to maintain albumin levels above 30 g/L during the postoperative period. The dose is similarly calculated based on the albumin deficit and patient weight.
  Arms: High Albumin Threshold Group (30 g/L)(HAT Group)

SUMMARY:
This study aims to evaluate the impact of goal-oriented albumin infusion on short-term postoperative outcomes in gastric cancer patients. It is a single-center, prospective, non-randomized controlled study. Patients are divided into two groups: the experimental group receives albumin infusion when serum albumin levels fall below 25 g/L, while the control group receives albumin infusion when levels fall below 30 g/L. The primary endpoint is the incidence of complications graded Clavien-Dindo III or above within 30 days post-surgery. Secondary endpoints include nutritional recovery, gastrointestinal function recovery, hospital stay duration, and overall complication rates. The study seeks to optimize perioperative albumin management strategies and improve clinical outcomes.

DETAILED DESCRIPTION:
Detailed Description:

This study evaluates the application and impact of goal-oriented albumin infusion in managing postoperative complications in gastric cancer patients. It is designed as a single-center, prospective, non-randomized controlled trial. The study population includes adult patients (18-80 years) undergoing radical gastric cancer surgery. Patients are divided into two groups:

Experimental Group: Albumin infusion is initiated when serum albumin levels fall below 25 g/L, aiming to maintain levels above this threshold.

Control Group: Albumin infusion is initiated when serum albumin levels fall below 30 g/L, maintaining levels above this threshold.

The primary endpoint is the incidence of complications graded Clavien-Dindo III or above within 30 days postoperatively. Secondary endpoints include nutritional status recovery (albumin levels within the first 7 days), hospital stay duration, gastrointestinal recovery (first flatus and bowel movement), and overall complication rates.

This study dynamically monitors albumin levels and evaluates the effects of different infusion standards on short-term postoperative outcomes. By analyzing these outcomes, the research aims to provide evidence-based recommendations for optimizing perioperative albumin management strategies in gastric cancer patients.

Albumin infusions are conducted following established protocols, with dosage calculated based on the patient's serum albumin levels and weight. Strict inclusion and exclusion criteria ensure participant safety and study validity. Adverse events are monitored closely, and any serious events are reported to the ethics committee promptly.

Data will be collected using electronic case report forms (eCRFs) and analyzed using appropriate statistical methods, including propensity score matching and multivariable regression, to control for potential confounding factors. The study's findings will contribute to improving postoperative care in gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18 to 80 years old, suitable for patients undergoing gastric cancer surgery.
2. Gastric cancer diagnosis: gastric cancer patients confirmed by pathology, regardless of pathological type.
3. Cancer staging: Patients with preoperative CT assessment of TNM stage I to III and undergoing laparoscopic gastric cancer surgery or open gastric cancer surgery can be included.
4. Preoperative nutritional status: serum albumin level ≥ 30g/L, NRS-2002 score ≤ 2.
5. Type of surgery: patients who undergo any radical gastric cancer surgery (no restriction on surgical type, covering partial gastrectomy, total gastrectomy, etc.).
6. The patient gave informed consent to this study and signed the corresponding informed consent form.
7. ASA classification I-III.
8. ECOG score ≤ 2

Exclusion Criteria:

1. Preoperative acute infection: Acute infection or acute complications (such as pneumonia, urinary tract infection, gastrointestinal bleeding, perforation, obstruction, etc.) have been diagnosed before surgery.
2. Immunosuppressed patients: such as long-term use of immunosuppressants (such as glucocorticoids), organ transplant patients, or those who have been diagnosed with HIV infection.
3. Serious basic diseases: such as severe liver insufficiency (Child Pugh class B or C), renal insufficiency (serum creatinine>133umol/L), severe cardiac insufficiency (NYHA class III and above), severe pulmonary insufficiency (preoperative blood gas analysis PaO2 ≤ 60mmHg).
4. Patients with a history of albumin allergy.
5. Intraoperative blood loss is greater than 500ml.
6. Preoperative hemoglobin <70g/L.
7. Receive neoadjuvant radiotherapy before surgery.
8. Patients who require combined organ resection.
9. Patients who are found to have distant metastasis during intraoperative exploration, or who can not undergo radical resection.

Withdrawal Criteria:

1) During the trial, the subjects suffered severe allergic reactions due to albumin infusion, such as acute anaphylactic shock, airway edema, hypotension, etc., and were not suitable for continued use of albumin. 2) If the subject clearly expresses his unwillingness to continue participating in the experiment due to personal reasons, even if his physical condition allows continued intervention, respect the patient's wishes and terminate his participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Complications (Clavien-Dindo Grade III or Above) | 30 Days Post-Surgery
  The primary outcome measure is the incidence of severe postoperative complications graded as Clavien-Dindo Grade III or above. These complications include those requiring surgical, endoscopic, or radiological intervention, or resulting in life-threatening conditions or mortality. The measure aims to compare the effects of two different albumin infusion thresholds (25 g/L vs. 30 g/L) on the rate of severe complications within the study period.

SECONDARY OUTCOMES:
Serum Albumin Levels Post-Surgery | 7 Days Post-Surgery
  The change in serum albumin levels within the first 7 days post-surgery will be measured to assess the effectiveness of goal-oriented albumin infusion in maintaining adequate protein levels. This measure will help evaluate nutritional recovery and the physiological impact of the intervention.
Length of Hospital Stay | From the day of surgery to the day of discharge (up to 30days)
  Postoperative length of hospital stay, measured in days from the day of surgery to the day of discharge.
Gastrointestinal Recovery | Postoperative Day 1 to Day of Discharge (approximately Day 7）
  The time to first flatus and bowel movement after surgery will be measured from postoperative day 1 to the day of discharge, to evaluate the recovery of gastrointestinal function and the influence of different albumin thresholds on postoperative recovery.
Overall Postoperative Complication Rate | 30 Days Post-Surgery
  The overall rate of postoperative complications, including all Clavien-Dindo grades (I to V), will be recorded and analyzed. This measure aims to assess the broader impact of goal-oriented albumin infusion on postoperative outcomes across all severity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Yuchen Guo, Ph.D., Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
If other researchers can provide valid reasons or demonstrate a need for additional collaboration, we may consider to share the data upon their request after we complete our study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after we complete our study.
Access Criteria: Researchers can provide valid reasons or demonstrate a need for additional collaboration with us.